CLINICAL TRIAL: NCT01269294
Title: A Double-blind, Double-dummy, Randomized, 4-period Cross-over, Placebo- and Positive-controlled Study to Evaluate the Effect of TMC435 on the QTc Interval in Healthy Subjects
Brief Title: TMC435-TiDP16-C117: The Effect of TMC435 on the Results of Electrocardiograms (Electric Recording of the Heart) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017491; TMC435-TiDP16-C117 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2010-12-30; First posted 2011-01-04 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435-TiDP16-C117; TMC435-C117; TMC435; HCV; Moxifloxacin; ECG; QT; QTc
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 001 (Experimental): TMC435 2 capsules of 75 mg once daily for 7 days in Treatment A
  Interventions: Drug: TMC435
- 002 (Other): Placebo for TMC435 2 placebo capsules once daily for 7 days in Treatment A
  Interventions: Drug: Placebo for TMC435
- 003 (Other): Placebo for moxifloxacin 1 placebo tablet on Day 7 of Treatments A B and D
  Interventions: Drug: Placebo for moxifloxacin
- 004 (Experimental): TMC435 2 capsules of 75 mg and 2 capsules of 100 mg once daily for 7 days in Treatment B
  Interventions: Drug: TMC435
- 005 (Other): Placebo for TMC435 4 placebo capsules once daily for 7 days in Treatment C
  Interventions: Drug: Placebo for TMC435
- 006 (Other): Moxifloxacin 1 tablet of 400 mg on Day 7 of Treatment C
  Interventions: Drug: Moxifloxacin
- 007 (Placebo Comparator): Placebo for TMC435 4 placebo capsules once daily for 7 days in Treatment D
  Interventions: Drug: Placebo for TMC435

INTERVENTIONS:
Drug: TMC435 — 2 capsules of 75 mg once daily for 7 days in Treatment A
  Arms: 001
Drug: Placebo for TMC435 — 4 placebo capsules once daily for 7 days in Treatment C
  Arms: 005
Drug: TMC435 — 2 capsules of 75 mg and 2 capsules of 100 mg once daily for 7 days in Treatment B
  Arms: 004
Drug: Placebo for TMC435 — 2 placebo capsules once daily for 7 days in Treatment A
  Arms: 002
Drug: Moxifloxacin — 1 tablet of 400 mg on Day 7 of Treatment C
  Arms: 006
Drug: Placebo for moxifloxacin — 1 placebo tablet on Day 7 of Treatments A, B and D
  Arms: 003
Drug: Placebo for TMC435 — 4 placebo capsules once daily for 7 days in Treatment D
  Arms: 007

SUMMARY:
The purpose of this study is to evaluate the effect of TMC435 on the results of electrocardiograms (ECGs) in healthy volunteers. An electrocardiogram is an electric recording of the heart. TMC435 is being investigated for the treatment of chronic hepatitis C virus infection.

DETAILED DESCRIPTION:
This is a double-blind, double-dummy, randomized, 4-period cross-over, placebo- and positive-controlled, Phase I study. This means neither the study doctor nor the participants know in which treatment session you will receive which active medication or matching placebo. Every participant will receive 4 treatment sessions (Treatments A, B, C and D) in a different order. The order in which you receive the treatment sessions is determined by chance, like tossing a coin. The purpose of the study is to evaluate the effect of TMC435 on the results of electrocardiograms (electric recording of the heart). Two dose regimens of TMC435 will be tested, ie, 150 mg once daily (the dose that will be given to patients) and 350 mg once daily (a dose higher than the one that will be given to patients), administered for 7 days. A single dose of 400 mg moxifloxacin will be used as a positive control to assess trial sensitivity. The trial population will consist of 60 healthy volunteers of which approximately 18 will be females. In each treatment, dummy capsules will be added in order to have the same number of capsules in each treatment. Treatment A will consist of 150 mg TMC435 once daily for 7 days (2 capsules of TMC435 and 2 capsules placebo on days 1-7, 1 placebo tablet for moxifloxacin on Day 7). Treatment B will consist of 350 mg TMC435 once daily for 7 days (4 capsules of TMC435 on Days 1-7, 1 placebo tablet for moxifloxacin on Day 7). Treatment C will consist of 400 mg moxifloxacin on Day 7 (4 capsules of placebo for TMC435 on Days 1-7, 1 moxifloxacin tablet on Day 7). In Treatment D only placebo will be given (4 capsules of placebo for TMC435 on Days 1-7, 1 placebo tablet for moxifloxacin on Day 7). There will be a washout period of at least 10 days between subsequent treatments. A pharmacogenomic blood sample (DNA sample, blood sample from which your genetic information can be analyzed) will be collected from all volunteers and will be analyzed upon observation of irregular electrocardiogram during the study. The purpose is to see if irregularities in the electrocardiogram can be linked to genetic variants. DNA samples may also be analyzed for additional genes related to pharmacokinetics (what the body does with the drug), pharmacodynamics (what the drug does to your body) or safety and tolerability of TMC435 during the study, as necessary. Two oral doses of TMC435 (150 or 350 mg) or placebo will be given once daily for 7 consecutive days. A single dose of moxifloxacin 400 mg will be administered orally on Day 7 in one of the treatment sessions only.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers for at least six months
* Have a body mass index of 18.0 to 30.0 kg per square meter
* Be healthy on the basis of physical examination, medical history, vital signs, and clinical laboratory tests performed at screening.

Exclusion Criteria:

* Use of disallowed therapies, including over-the-counter products and dietary supplements
* Any skin condition likely to interfere with ECG electrode placement or adhesion
* History or evidence of current use of alcohol or recreational or narcotic drug use
* Clinically relevant abnormality on ECG at screening or history of clinically relevant heart rhythm disturbances.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in QT/QTc interval for TMC435 therapeutic dose versus placebo | 24-hour measurement on Day 7 of Treatment Session A and D
Change in QT/QTc interval for TMC435 supratherapeutic dose versus placebo | 24-hour measurement on Day 7 of Treatment Session B and D

SECONDARY OUTCOMES:
RR interval, HR, PR interval, QRS interval and ECG morphology | 1-hour predose measurement on Day 1 of every treatment session
RR interval, HR, PR interval, QRS interval and ECG morphology | 24-hour measurement on Day 7 of every treatment session
Pharmacokinetics of 150 mg TMC435 once daily for 7 days | Predose on Day 1 of every treatment and on Days 5 and 6 of Treatments A and B. 24 hour profile on Day 7 of Treatment A and B
Pharmacokinetics of 350 mg TMC435 once daily for 7 days | Predose on Day 1 of every treatment and on Days 5 and 6 of Treatments A and B. 24 hour profile on Day 7 of Treatment A and B
Changes from baseline for electrocardiogram (ECG) and physical examination | During all treatment sessions: Daily safety ECG from Day -1 to Day 9 with on Day 1 and 7 an additional safety ECG at 5h timepoint plus at screening and follow-up visits. Physical examination at screening, on Day 8 and at the follow-up visits
Number of participants with adverse events and severity of adverse events | From signing of informed consent onwards until last trial-related visit
Changes from baseline and percentage of subjects with abnormal values for laboratory parameters | At screening, on Days -1, 1, 5, 8 of all treatment sessions and at the follow-up visits
Changes from baseline and percentage of subjects with abnormal values for pulse and blood pressure | At screening, daily from Day -1 to Day 9 with a second measurement on Day 7 of all treatment sessions and at the follow-up visits
Difference of QTc between moxifloxacin treatment and placebo treatment as a measure for trial sensitivity | On Day 7 of Treatment C and D, at the 2, 3, 4 and 5 hour timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited